CLINICAL TRIAL: NCT06603155
Title: Phase 2, Single Arm Study to Evaluate the Efficacy of Time Restricted Eating (TRE) on Immunotherapy Treatment Outcomes in Patients With Metastatic Head and Neck Squamous Cell Cancer (mHNSCC) or Unresectable or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Time Restricted Eating (TRE) in Metastatic Head and Neck Squamous Cell Cancer (mHNSCC) or Unresectable or Metastatic Renal Cell Carcinoma (RCC)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changing priorities of portfolio
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00115641
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Head-and-neck Squamous-cell Carcinoma; Unresectable Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (TRE) for mHNSCC participants (Experimental)
  Interventions: Behavioral: Time restricted eating (TRE)
- Time Restricted Eating (TRE) for RCC participants (Experimental)
  Interventions: Behavioral: Time restricted eating (TRE)

INTERVENTIONS:
Behavioral: Time restricted eating (TRE) — TRE is defined as limiting daily food intake to 10 hour period with a nightly fasting period of 14 hours.

SUMMARY:
The purpose of this study is to evaluate whether Time Restricted Eating (TRE) can improve responses in participants with metastatic head and neck squamous cell cancer (mHNSCC) or unresectable/metastatic renal cell carcinoma (RCC) receiving Immune Checkpoint Blockers (ICB) by changing the gut microbiome (the bacteria and other microorganisms living in individual's bodies). A particular focus of this study is to compare the outcomes of African American participants when compared to the rest of the participant population. TRE is a form of intermittent fasting where food and drink intake is limited to a specific time window during the day. The information learned from this study may help researchers develop new strategies to improve outcomes in patients with mHNSCC and RCC in the future.

Participants will be asked to complete a dietary survey at baseline and week 9 and provide a baseline stool and blood sample. Two weeks before beginning ICB and after participants completed the baseline assessments, they will begin TRE. TRE will be defined as limiting food and drink intake to a 10 hour window during each day and fasting for 14 hours at night. Participants will be asked to complete a daily food log to document the times they eat and drink. On day 1 of ICB and weeks 3, 6, 9, 26, and 52 after ICB, participants will be asked to collect a blood sample and a toxicity assessment will be performed. On day 1 of ICB and weeks 9, 26, and 52 of ICB, participants will be asked to provide a stool sample. Participants will also undergo tumor imaging throughout the study as part of their standard of care assessments. If a participant's disease progresses after ICB, they will repeat all study assessments and be withdrawn from the study.

ELIGIBILITY:
HNSCC Cohort

Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent/metastatic head and neck squamous cell cancer that is not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy) and initiating standard of care immune checkpoint blocker- (Nivolumab, pembrolizumab, Atezolizumab, Avelumab or Durvalumab with or without chemotherapy), for the first time.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
4. Age ≥18 years, able to understand and voluntarily consent.

Exclusion Criteria:

1. BMI < 18.5.
2. Diabetes mellitus, pregnancy, any eating disorder including anorexia nervosa or bulimia.
3. Ongoing or active infection requiring iv antibiotics, autoimmune disease requiring systemic steroids greater than prednisone 60 mg equivalent, symptomatic congestive heart failure, unstable angina pectoris, insulin use, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients who have known leptomeningeal metastases or untreated or symptomatic brain metastases. Eligible patients must be neurologically asymptomatic and not requiring steroids.
5. Has received prior therapy with any anti-PD-1, anti-PDL-1 in a metastatic setting.
6. Patients for whom fasting is medically contraindicated

RCC Cohort

Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable/metastatic clear cell renal cell carcinoma that is not amenable to local therapy with curative intent (surgery, radiation therapy, cryoablation, etc.,) and initiating standard of care systemic therapy consisting of immune checkpoint blockade (e.g. ipilimumab/nivolumab, cabozantinib/nivolumab, lenvatinib/pembrolizumab, or axitinib/pembrolizumab) for the first time.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
4. Age ≥18 years, able to understand and voluntarily consent.

Exclusion Criteria:

1. BMI < 18.5.
2. Diabetes mellitus, pregnancy, any eating disorder including anorexia nervosa or bulimia.
3. Ongoing or active infection requiring iv antibiotics, autoimmune disease requiring systemic steroids greater than prednisone 60 mg equivalent, symptomatic congestive heart failure, unstable angina pectoris, insulin use, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients who have known leptomeningeal metastases or untreated or symptomatic brain metastases. Eligible patients must be neurologically asymptomatic and not requiring steroids.
5. Has received prior therapy with any anti-PD-1, anti-PDL-1
6. Patients for whom fasting is medically contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival (PFS) for HNSCC cohort only | 1 Year
  Time from enrollment to radiographic disease progression as per RECIST 1.1 or death from any cause
Time restricted eating (TRE) associated change in gut microbiome | Baseline, Day 1, Week 9, Week 26 and Week 52
  Microbiome changes in stool
Time restricted eating (TRE) associated change in metabolome | Baseline, Day 1, Week 9, Week 26 and Week 52
  Metabolomics in blood
Time restricted eating (TRE) associated change in IGF1 | Baseline, Day 1, Week 9, Week 26 and Week 52
  IGF1 level in blood
Time restricted eating (TRE) associated change in immune repertoire | Baseline, Day 1, Week 9, Week 26 and Week 52
  Comprehensive analysis of effector T cells and suppressor T cell populations in PBMC, plasma cytokines will be carried out
Response to immune checkpoint blocker (ICB) at first response assessment | Week 9
  Radiographic response as per RECIST 1.1

SECONDARY OUTCOMES:
1-year immune related adverse events (irAE) rate | 1 Year
  1 year rate of irAE, as per CTCAE v.5
Feasibility of Time restricted eating (TRE) in African American HNSCC participants on immune checkpoint blocker (ICB) | Through Week 52
  Number of African American participants who were compliant, which is defined as 14 hr TRE daily for 5 days per week, for 9 out of first 12 weeks (70%)
1-year immune related adverse events (irAE) rate in African American participants | 1 year
  1 year rate of irAE, as per CTCAE v.5 in African American participants
Median progression free survival (PFS) for RCC cohort only | 1 Year
  Time from enrollment to radiographic disease progression as per RECIST 1.1 or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No